CLINICAL TRIAL: NCT01017081
Title: Chest Physiotherapy in Pediatric Patients Hospitalised With Community-acquired Pneumonia: a Randomized Clinical Trial
Brief Title: Chest Physiotherapy in Pediatrics Patients With Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santa Casa de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Universidade Federal do Rio Grande do Sul, Janice Luisa Lukrafka
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FISIOPUL
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Pneumonia
Keywords: physiotherapy; children; clinical trial
MeSH Terms: conditions — Pneumonia | interventions — Physical Therapy Modalities; Patient Positioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Non-mandatory request to maintain lateral positioning to improve air exchange, to cough in order to clear secretion, and to perform diaphragmatic and deep breathing, for five minutes, once a day, during hospital stay.
  Interventions: Other: Positioning and cough
- Physiotherapy (Experimental): Physiotherapy: Children younger than 5 years: Manual Thoracic vibration (TV), thoracic compression (TC), positive expiratory pressure (PEP), and forced exhalation with the glottis open ("huffing"). Children aged 5 years or older: same procedures in addition to the ventilatory patterns, and a forced expiratory technique (FET), consisting of one or two "huffs" (forced expirations) followed by a period of relaxed, controlled diaphragmatic breathing, three times per day, for 10 to 12 minutes, during hospital admission.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy: three times per day, for 10 to 12 minutes, during hospital admission
  Arms: Physiotherapy
Other: Positioning and cough — Non-mandatory request to maintain lateral positioning to improve air exchange and cough
  Arms: Control

SUMMARY:
Chest physiotherapy has been used to treat pediatric patients hospitalized with pneumonia however there was no evidence to support a beneficial effect in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 12 years with acute community-acquired pneumonia (cough, tachypnea, fever and with a chest radiography with lobar, segmental or bronchopneumonia within the first 48 hours)

Exclusion Criteria:

* Severely ill patients (hospitalized in intensive care units)
* Pleural effusion treated with chest drainage
* Atelectasis detected by x-ray
* Pneumonia or pleural effusion in the previous six months
* Other pulmonary underlying disease, heart disease, cerebral palsy or immune deficiency

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2001-09; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa de Porto Alegre, Posto Alegre, Rio Grande do Sul, Brazil